CLINICAL TRIAL: NCT05580965
Title: The Effect of Duration of Pressure Applied After Blood Sample Collection on the Development of Ecchymosis in Geriatric Patients Using Oral and Subcutaneous Anticoagulants: A Randomized Controlled Trial
Brief Title: Blood Sample Collection in Geriatric Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Tulay Basak, Professor, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 779
Record Dates: First submitted 2022-10-07; First posted 2022-10-14 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Venipuncture Site Bruise

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- control group (No Intervention): Routine procedure
- Group A (Experimental): 1 min pressure applied
  Interventions: Other: 20 N pressure for 1 minute
- Group B (Experimental): 3 min pressure applied
  Interventions: Other: 20 N pressure for 3 minute
- Group C (Experimental): 5 min pressure applied
  Interventions: Other: 20 N pressure for 5 minute

INTERVENTIONS:
Other: 20 N pressure for 1 minute — After blood collection, 20 N pressure applied for 1 minute
  Arms: Group A
Other: 20 N pressure for 3 minute — After blood collection, 20 N pressure applied for 3 minute
  Arms: Group B
Other: 20 N pressure for 5 minute — After blood collection, 20 N pressure applied for 5 minute
  Arms: Group C

SUMMARY:
This study aimed to evaluate the effect of different durations of a specific pressure applied after blood collection on the development of ecchymosis in geriatric patients using oral and subcutaneous anticoagulants.

DETAILED DESCRIPTION:
The research sample consisted of patients hospitalized in the Geriatrics Clinic of a city hospital. This study aimed to evaluate the effect of different durations of a specific pressure applied after blood collection on the development of ecchymosis in geriatric patients using oral and subcutaneous anticoagulants. In this study, whether ecchymosis developed at the 24th, 48th and 72nd hours after the blood collection procedure was evaluated.

ELIGIBILITY:
Inclusion Criteria:

* patients aged 65 years and over
* who voluntarily agreed to participate in the study
* who used oral (Rivaroxaban 10-15-20 mg, Dabigatran, 75-110-150 mg, Apixaban 2.5-5 mg) and subcutaneous (Enoxaparin sodium 6000-4000 anti-Xa IU/0.6-0.4 ml) anticoagulants
* who were literate in Turkish
* who were scheduled for blood collection
* who would undergo blood collection from the antecubital site with vacutainer

Exclusion Criteria:

* patients with communication problems
* patients with hematoma, ecchymosis, and scarring in the antecubital site
* patients who would be discharged before 72 hours
* patients with coagulation disorders

Ages: 65 Years to 93 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 164 (Actual)
Dates: Start 2021-10-30 (Actual); Primary Completion 2022-06-15 (Actual); Study Completion 2022-06-15 (Actual)

PRIMARY OUTCOMES:
number of participants with ecchymosis developed. | at the 24 th hours
  In this study, whether ecchymosis developed at the 24th, 48th, and 72nd hours after the blood collection procedure was evaluated.
number of participants with ecchymosis developed. | at the 48 th hours
  In this study, whether ecchymosis developed at the 24th, 48th, and 72nd hours after the blood collection procedure was evaluated.
number of participants with ecchymosis developed. | at the 72 nd hours
  In this study, whether ecchymosis developed at the 24th, 48th, and 72nd hours after the blood collection procedure was evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Tülay Başak, Principal Investigator — Saglik Bilimleri Universitesi
Locations (1):
- Tulay Basak, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No